CLINICAL TRIAL: NCT01793077
Title: Phase IV, Non-interventional, Prospective, Open Label, Non Comparative Real Life Data Collection of Depo-Eligard® 7.5 mg, 22.5 mg and 45 mg in Male Prostate Cancer Patients
Brief Title: Observational, Non-interventional, Non Comparative Real Life Data Collection of Depo-Eligard® 7.5 mg, 22.5 mg and 45 mg in Male Prostate Cancer Patients
Acronym: TREMODI
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Veeda Clinical Research (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: BE-11-EGD-04
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Phase 4; Data collection; Observational; Depo-Eligard; Prospective; Non-interventional; Treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate Cancer patients
  Interventions: Drug: Depo-Eligard®

INTERVENTIONS:
Drug: Depo-Eligard® — Subcutaneous
  Other Names: Leuprolide Acetate

SUMMARY:
Tremodi is an observational, non-interventional, prospective, open-label, non-comparative study that will collect real life data of a treatment with Depo-Eligard® in 3 different administrations in male prostate cancer patients.

Once the examining physician has decided on the therapeutic approach and if the selection criteria are fulfilled, he will propose the patient to participate in the study. An informed consent form will be collected for all participants in the study.

There are 2 possible study visits that coincide with a routine consultation, namely visit 1 (inclusion visit) and visit 2 (end of study visit). On both visits, Adverse Drug Reactions (adverse event caused by Depo-Eligard®) are collected and the patient will be asked to complete a Quality Of Life questionnaire (EORTC QLQ-C30). At visit 2, the examining physician will give a global evaluation of the treatment with Depo-Eligard® and assesses the treatment benefit of the patient.

Testosterone and Prostate Specific Antigen (PSA) blood values are collected during both visits, if available.

ELIGIBILITY:
Inclusion Criteria:

* Patients having been prescribed Depo-Eligard® 7.5 mg - 22.5 mg - 45 mg in accordance with the terms of the marketing authorization.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consultation at urology department
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of tolerability of treatment on a 4 point scale | Last Visit (after at least 180 days of treatment)

SECONDARY OUTCOMES:
Occurrence of Adverse Drug Reactions | Day 1 and Last Visit (after at least 180 days of treatment)
Investigator satisfaction with treatment | Last Visit (after at least 180 days of treatment)
Overall patient's assessment of treatment benefit | Last Visit (after at least 180 days of treatment)
Changes in quality of life of subjects as measured by EORTC QLQ-C30 | Day 1 and Last Visit (after at least 180 days of treatment)
  European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-C 30 (EORTC-QLQ-C30)
Frequency of use of dosing schedules of Depo-Eligard® and the reasons for selecting a schedule | Day 1 and Last Visit (after at least 180 days of treatment)
Efficacy of treatment | Day 1 and Last Visit (after at least 180 days of treatment)
  (1) Changes in PSA and testosterone levels if available, (2) Change in disease symptoms and (3) Objective disease response

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (23):
- Belgium (23):
  - Site: 5, Antwerp, Antwerp
  - Site: 8, Antwerp, Antwerp
  - Site: 9, Antwerp, Antwerp
  - Site: 14, Antwerp, Antwerp
  - Site: 4, Antwerp, Antwerp
  - Site: 33, Merksem, Antwerp
  - Site: 1, Turnhout, Antwerp
  - Site: 23, Brussels, Brussels Capital
  - Site: 13, Brussels, Brussels Capital
  - Site: 24, Uccle, Brussels Capital
  - Site: 32, Aalst, East Flanders
  - Site: 34, Dendermonde, East Flanders
  - Site: 11, Ghent, East Flanders
  - Site: 17, Oudenaarde, East Flanders
  - Site: 18, Tienen, Flemish Brabant
  - Site: 39, La Louvière, Hainaut
  - Site: 37, Sint-Truiden, Limburg
  - Site: 38, Liège, Liège
  - Site: 26, Lasne-Chapelle-Saint-Lambert, Walloon Brabant
  - Site: 21, Ieper, West Flanders
  - Site: 20, Izegem, West Flanders
  - Site: 25, Kortijk, West Flanders
  - Site: 31, Ostend, West Flanders